CLINICAL TRIAL: NCT05192954
Title: Comparing Postoperative Pain After LigaSureTM Vessel Sealing Device Versus Conventional Suturing Methods for Vaginal Hysterectomy and Pelvic Reconstructive Surgery: a Randomized Controlled Trial
Brief Title: Comparing Postoperative Pain After Vessel Sealing Device Versus Conventional Suturing Methods for Vaginal Hysterectomy and Pelvic Reconstructive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marlana McDowell (Other)
Collaborators: TriHealth Hatton Research Institute (Other)
Responsible Party: Sponsor-Investigator, Marlana McDowell, Female Pelvic Medicine and Reconstructive Surgery Fellow, TriHealth Inc.
Organization: TriHealth Inc. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-094
Record Dates: First submitted 2021-12-29; First posted 2022-01-14 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; Vaginal Hysterectomy; Vaginal Vault Suspension; Prolapse Repair
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: Single-blinded randomized controlled trial
Who Masked: Participant
Masking Description: Participant will be under anesthesia and will not know which surgical method is being utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vessel sealing device (Experimental): Vessel sealing device to be utilized for vaginal hysterectomy
  Interventions: Device: LigaSureTM vessel sealing device
- Conventional clamping and suturing method (No Intervention): Vaginal hysterectomy will be performed utilizing conventional Heaney clamps, scissors, and suturing material.

INTERVENTIONS:
Device: LigaSureTM vessel sealing device — Device will be used to clamp, cauterize, seal, and transect tissue during vaginal hysterectomy.
  Other Names: LigaSure; LigaSureTM; Electrosurgical sealing device
  Arms: Vessel sealing device

SUMMARY:
This study will investigate pain outcomes for patients undergoing vaginal hysterectomy with pelvic reconstructive surgery using the LigasureTM vessel sealing device as compared to conventional clamping and suturing methods.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, able to understand informed consent
* Vaginal hysterectomy with vaginal vault suspension
* with or without anterior and posterior repairs
* with or without removal of fallopian tubes or ovaries
* with or without procedures for stress urinary incontinence

Exclusion Criteria:

* Use of mesh for prolapse repair
* Robotic, laparoscopic, or open technique used for prolapse repair and/or hysterectomy
* Concomitant procedure done by an additional surgeon
* Concomitant anal sphincteroplasty or rectovaginal fistula repair
* History of chronic pelvic pain receiving medical care
* Daily use of medication for pain: NSAID, Tylenol, opioid, gabapentin, and/or amitriptyline
* Pregnancy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 3-6 hours postoperative
  Visual Analog Scale, 0-10, with 10 being "most severe pain"

SECONDARY OUTCOMES:
Vaginal Pain | 3-6 hours postoperative
  Visual Analog Scale, 0-10, with 10 being "most severe pain"
Abdominal Pain | 3-6 hours postoperative
  Visual Analog Scale, 0-10, with 10 being "most severe pain"

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Yeung, DO, Principal Investigator — TriHealth Inc.
Locations (2):
- United States (2):
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ray MM, Crisp CC, Pauls RN, Hoehn J, Lewis K, Bonglack M, Yeung J. Use of a Vessel Sealer for Hysterectomy at Time of Prolapse Repair: A Randomized Clinical Trial. Urogynecology (Phila). 2025 Mar 1;31(3):234-242. doi: 10.1097/SPV.0000000000001617. Epub 2024 Dec 9. PMID 39657205